CLINICAL TRIAL: NCT01991470
Title: A Performance Evaluation of the Enlite™ and Enlite 3 Glucose Sensor to Support Use in Children
Brief Title: CEP249 Pediatric Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CEP249
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Insulin Requiring Diabetes
Keywords: Insulin requiring diabetes; Children; Sensor; Accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enlite sensors (Experimental): Each subject will first wear enlite sensors and will come for clinic visit for YSI (Yellow Spring Instruments). Then each subject will wear enlite 3 sensors and will come for clinic visit for YSI (Yellow Spring Instruments) or SMBG (Self-Monitoring of Blood Glucose) testing. SMBG testings are for subjects 2-6 years of age and cannot tolerate YSI. In addition. In addition, subjects aged 2-6 years old will not participate in Enlite phase. They only participate in Enlite 3 phase.
  Interventions: Device: Enlite sensors

INTERVENTIONS:
Device: Enlite sensors — Subject wears enlite sensor first and followed by enlite 3 sensor.

SUMMARY:
The purpose of this study is to evaluate the Enlite Sensor™ and Enlite 3 Sensor performance in pediatric patients with insulin requiring diabetes at the beginning, middle and end of sensor wear.

DETAILED DESCRIPTION:
This study is a prospective, single arm, multi-center, in-clinic study.. There will be two consecutive phases of the study:

A total of up to 260 subjects (2-18 years old) will be enrolled at up to 15 investigational centers

Subjects will come for clinic visit for YSI reference glucose testing and for Enlite Sensor™ and Enlite 3 Sensor™ testing. SMBG (Self-Monitoring of Blood Glucose) reference measurement is for subjects 2-6 years of age and cannot tolerate YSI.

Study has a run-in period and a study period with a total of 10 visits

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 2-18 years of age at time of screening
2. Subject has been diagnosed with insulin requiring diabetes mellitus for at least one year.
3. Subject is willing to perform greater than or equal to 4 finger stick blood glucose measurements daily
4. Subject is willing to perform required sensor calibrations
5. Subject is willing to wear the system (Guardian Mobile application, pumps, sensors, meter) continuously throughout the study
6. Adequate venous access as assessed by investigator or appropriate staff

Exclusion Criteria:

1. Subject is unable to tolerate tape adhesive in the area of sensor placement
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Females of child-bearing potential who have a positive pregnancy test at screening or plans to become pregnant during the course of the study
5. Subjects with hematocrit lower than the normal age specific reference range per central or local lab testing

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brazg, MD, Principal Investigator — Rainier Clinical Research Center; Timothy Bailey, MD, Principal Investigator — AMCR Institute; Jeanie Tryggestad, MD, Principal Investigator — OUHSC Department of Pediatrics; Linda DiMeglio, MD, Principal Investigator — Indiana University, Riley Hospital for Children; Larry Fox, MD, Principal Investigator — Nemours Children's Clinic; Jennifer Sherr, MD, Principal Investigator — Yale University, Yale Diabetes Research Program; Robert Slover, MD, Principal Investigator — Barbara Davis Center; Eva Tsalikian, MD, Principal Investigator — University of Iowa Children Hospital; Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Kevin Kaiserman, MD, Principal Investigator — SoCal Diabetes; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (11):
- United States (11):
  - AMCR Institute, Escondido, California
  - SoCal Diabetes, Torrance, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, Yale Diabetes Research Program, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - "Atlanta Diabetes Associates, Atlanta, Georgia
  - Indiana University, Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Children Hospital, Iowa City, Iowa
  - OUHSC Department of Pediatrics, Oklahoma City, Oklahoma
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Slover RH, Tryggestad JB, DiMeglio LA, Fox LA, Bode BW, Bailey TS, Brazg R, Christiansen MP, Sherr JL, Tsalikian E, Kaiserman KB, Sullivan A, Huang S, Shin J, Lee SW, Kaufman FR. Accuracy of a Fourth-Generation Continuous Glucose Monitoring System in Children and Adolescents with Type 1 Diabetes. Diabetes Technol Ther. 2018 Sep;20(9):576-584. doi: 10.1089/dia.2018.0109. Epub 2018 Jul 31. PMID 30063162

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two phase study: Enlite and Enlite 3. Some participated only Enlite phase and some only participated in Enlite 3 phase.
Groups:
- 2-18 Years Old Wearing Sensors: 2-18 years old wearing Enlite and/or Enlite3 sensors.
Period: Enlite 1 Period
Arm/Group | 2-18 Years Old Wearing Sensors
Started | 161
Completed | 141
Not Completed | 20
Not completed — Withdrawal by Subject | 18
Not completed — Adverse Event | 1
Not completed — Inclusion/Exclusion not met | 1
Period: Enlite 3 Period
Arm/Group | 2-18 Years Old Wearing Sensors
Started | 158 (Additional 25 subjects who participated only Enlite 3 phase)
Completed | 146
Not Completed | 12
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Physician Decision | 8
Not completed — DUE TO MULTIPLE SENSOR ISSUES | 1

BASELINE CHARACTERISTICS:
Population: a total of 186 subjects participated the study
Groups:
- 2-18 Year Olds Wearing Enlite Sensor: 2-18 years old wearing Enlite and/or Enlite3 sensors.
Arm/Group | 2-18 Year Olds Wearing Enlite Sensor
Number analyzed (Participants) | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 103
Region of Enrollment [Number; unit: participants]
  United States | 186

OUTCOME MEASURES:

1. Primary Outcome: Enlite Sensor Accuracy Mean Absolute Relative Difference (MARD), With Lower Serial Number 530G Pump
Description: Enlite Sensor accuracy relative to the YSI (Yellow Spring Instruments) reference. Each subject wore two 530G pumps. The results for the lower serial number pump worn by each subject were arbitrarily selected and pooled across subjects for the primary dataset. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days were pooled together for reporting purpose.
Time Frame: 6 days
Population: All subjects wearing Enlite sensor with lower serial number of 530G pump. A total of 30 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite Sensor Accuracy MARD, Lower Serial Number: Enlite Sensor accuracy relative to the YSI reference. Each subject wore two 530G pumps. The results for the lower serial number pump worn by each subject were arbitrarily selected and pooled across subjects for the primary dataset. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days were pooled together for reporting purpose.
Arm/Group | Enlite Sensor Accuracy MARD, Lower Serial Number
Number analyzed (Participants) | 131
percentage of difference | 15.02 (13.37)

2. Primary Outcome: Enlite 3 Sensor Accuracy Mean Absolute Relative Difference (MARD), With the Guardian Mobile System
Description: Enlite 3 Sensor accuracy using Guardian Mobile System compared to YSI or SMBG (Self-Monitoring of Blood Glucose) reference values. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 days
Population: a total of 25 subjects do not have device data
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite 3 Sensor Accuracy MARD, Guardian Mobile: Enlite 3 Sensor accuracy using Guardian Mobile System compared to YSI or SMBG reference values. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite 3 Sensor Accuracy MARD, Guardian Mobile
Number analyzed (Participants) | 133
percentage of difference | 10.88 (10.65)

3. Secondary Outcome: Enlite 3 Sensor Accuracy Mean Absolute Relative Difference (MARD), With the GST3C Transmitter
Description: Enlite 3 Sensor accuracy using GST3C transmitter used as a recorder compared to YSI or SMBG reference values. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 days
Population: A total of 41 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite 3 Sensor Accuracy MARD,GST 3C: Enlite 3 Sensor accuracy using GST3C transmitter used as a recorder compared to YSI or SMBG reference values. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite 3 Sensor Accuracy MARD,GST 3C
Number analyzed (Participants) | 117
percentage of difference | 11.08 (10.58)

4. Secondary Outcome: Enlite Sensor Accuracy Mean Absolute Relative Difference (MARD), With Higher Serial Number 530G Pump
Description: Enlite Sensor accuracy relative to the YSI reference. Each subject wore two 530G pumps. The results for the higher serial number pump worn by each subject were arbitrarily selected and pooled across subjects for the secondary dataset. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days were pooled together for reporting purpose.
Time Frame: 6 Days
Population: All subjects wearing Enlite sensors with high serial number 530G pump. A total of 35 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite Sensor Accuracy MARD, Higher Serial Number: Enlite Sensor accuracy relative to the YSI reference. Each subject wore two 530G pumps. The results for the higher serial number pump worn by each subject were arbitrarily selected and pooled across subjects for the secondary dataset. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days were pooled together for reporting purpose.
Arm/Group | Enlite Sensor Accuracy MARD, Higher Serial Number
Number analyzed (Participants) | 126
percentage of difference | 17.50 (19.70)

5. Secondary Outcome: Enlite Sensor Accuracy Mean Absolute Relative Difference (MARD), With Lower Serial Number 530G Pump, Using One Additional Calibration During FST
Description: Enlite Sensor accuracy relative to the YSI reference, using one additional calibration during FST. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days were pooled together for reporting purpose.
Time Frame: 6 Days
Population: A total of 32 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite Sensor Accuracy MARD, Lower Serial Number: Enlite Sensor accuracy using two 530G pumps and two REAL-Time transmitters with one additional calibration during FST will be evaluated and report separately (e.g., lower serial number and high serial number)Enlite sensor values will be compared to Yellow Spring Instruments (YSI) plasma glucose values during Frequent Sample Testing in the Enlite phase. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite Sensor Accuracy MARD, Lower Serial Number
Number analyzed (Participants) | 129
percentage of difference | 14.37 (12.99)

6. Secondary Outcome: Enlite Sensor Accuracy Mean Absolute Relative Difference (MARD), With Higher Serial Number 530G Pump, Using One Additional Calibration During FST
Description: as for outcome 5
Time Frame: 6 Days
Population: A total of 34 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite Sensor Accuracy MARD, Higher Serial Number: Enlite Sensor accuracy using two 530G pumps and two REAL-Time transmitters with one additional calibration during FST will be evaluated and report separately (e.g., lower serial number and high serial number) Enlite sensor values will be compared to Yellow Spring Instruments (YSI) plasma glucose values during Frequent Sample Testing in the Enlite phase. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite Sensor Accuracy MARD, Higher Serial Number
Number analyzed (Participants) | 127
percentage of difference | 16.94 (18.74)

7. Secondary Outcome: Enlite 3 Sensor Accuracy Mean Absolute Relative Difference (MARD), With the Guardian Mobile System, Using One Additional Calibration During FST
Description: Enlite 3 Sensor accuracy using Guardian Mobile System compared to YSI or SMBG reference values, with one additional calibration during FST. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 Days
Population: A total of 34 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite 3 MARD, Guardian Mobile, One Additional Fingerstick: Enlite 3 Sensor accuracy using, (1) Guardian Mobile System (2) GST 3C transmitter, with one additional calibration during FST will be evaluated and report. Enlite 3 sensor values will be compared to Yellow Spring Instruments (YSI) plasma glucose values during Frequent Sample Testing in the Enlite 3 phase. For subjects 2-6 years of age, SMBG may be used as a reference value. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite 3 MARD, Guardian Mobile, One Additional Fingerstick
Number analyzed (Participants) | 124
percentage of difference | 10.05 (9.26)

8. Secondary Outcome: Enlite 3 Sensor Accuracy Mean Absolute Relative Difference (MARD), With GST3C Transmitter, Using One Additional Calibration During FST
Description: Enlite 3 Sensor accuracy using GST3C transmitter used as a recorder compared to YSI or SMBG reference values, with one additional calibration during FST. For subjects 2-6 years of age, SMBG was used as a reference value if YSI cannot be tolerated. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Therefore, the unit of MARD is percentage (%). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 Days
Population: A total of 41 subjects did not have device data.
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- Enlite 3 MARD,GST 3C, One Additional Fingerstick: Enlite 3 Sensor accuracy using, (1) Guardian Mobile System (2) GST 3C transmitter, with one additional calibration during FST will be evaluated and report. Enlite 3 sensor values will be compared to Yellow Spring Instruments (YSI) plasma glucose values during Frequent Sample Testing in the Enlite 3 phase. For subjects 2-6 years of age, SMBG may be used as a reference value. MARD = Mean of ((Absolute difference of reference and Sensor glucose values / reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Arm/Group | Enlite 3 MARD,GST 3C, One Additional Fingerstick
Number analyzed (Participants) | 117
percentage of difference | 10.85 (10.35)

ADVERSE EVENTS:
Groups:
- 2-18 Year Olds Wearing Enlite Sensors: 2-18 year olds wearing Enlite Sensors
- 2-18 Year Olds Wearing Enlite3 Sensors: 2-18 year olds wearing Enlite3 Sensors
Arm/Group | 2-18 Year Olds Wearing Enlite Sensors | 2-18 Year Olds Wearing Enlite3 Sensors
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/158
Serious Adverse Events (participants affected / at risk) | 2/161 | 1/158
Other Adverse Events (participants affected / at risk) | 25/161 | 23/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-18 Year Olds Wearing Enlite Sensors (N=161) | 2-18 Year Olds Wearing Enlite3 Sensors (N=158)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pilonidal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Influenzavirus B (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-18 Year Olds Wearing Enlite Sensors (N=161) | 2-18 Year Olds Wearing Enlite3 Sensors (N=158)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Broken right thumb (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flu symptoms (Infections and infestations) | 1 (1) | 0 (0)
Food poisoning. (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypoglycemic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Insertion site pain (General disorders) | 1 (1) | 0 (0)
Laceration above right knee cap - requiring 9 sutures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left Broken Great Toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Puncture Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 1 (1) | 1 (1)
Stomach Virus (Infections and infestations) | 1 (1) | 0 (0)
Toe Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Resiratory Infection (Infections and infestations) | 3 (3) | 4 (4)
common cold (Infections and infestations) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
jaw pain due to wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0)
lowgrade fever, maximum 100.8 degrees (General disorders) | 1 (1) | 0 (0)
severe hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
vasovagal response (Nervous system disorders) | 1 (2) | 0 (0)
Abrasion on right arm and right leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cold sore (Infections and infestations) | 0 (0) | 1 (1)
Food Allergy: Shellfish Positive FPIES (Food PRotein Induced Enterocolitis Syndrome) (Immune system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Staff Infection left upper arm (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
hand, foot, mouth disease 0 (Infections and infestations) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sprain of left wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
vasovagal event (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No